CLINICAL TRIAL: NCT01015105
Title: Troponin Elevation in Consecutive Patients With Hip Fracture
Status: Completed | Type: Observational
Sponsor: Turku University Hospital (Other Government)
Responsible Party: Principal Investigator, Marjatta Strandberg, MD, Turku University Hospital
Other Study IDs: TnT in Hip Fracture
Record Dates: First submitted 2009-11-17; First posted 2009-11-18 (Estimated); Last update posted 2016-11-08 (Estimated); Status verified 2016-11

CONDITIONS: Hip Fracture
Keywords: patients with hip fracture
MeSH Terms: conditions — Hip Fractures | interventions — Observation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- patients with hip fracture
  Interventions: Other: observation

INTERVENTIONS:
Other: observation — observation

SUMMARY:
The aims of this study is to study the occurrence of the troponin elevations, ECG changes, and cardiac symptoms in unselected consecutive patients with hip fracture.

Followup will be carried out up to one year period.

ELIGIBILITY:
Inclusion Criterion:

* Hip fracture diagnosed in Turku Univeristy Hospital between October 2009 and May 2010

Exclusion Criterion:

* Patient refusal

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 200 patients with hip fracture
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2009-02; Primary Completion 2010-05 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Turku University Hospital, Turku, Finland

REFERENCES:
- [Derived] Nordling P, Kiviniemi T, Strandberg M, Strandberg N, Airaksinen J. Predicting the outcome of hip fracture patients by using N-terminal fragment of pro-B-type natriuretic peptide. BMJ Open. 2016 Feb 24;6(2):e009416. doi: 10.1136/bmjopen-2015-009416. PMID 26911583